CLINICAL TRIAL: NCT05335421
Title: The Influence of Mindfulness on Patient-Reported Outcomes Following Hip Preservation Surgery
Brief Title: Mindfulness and Hip Preservation Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0508; Protocol Version 10/13/2021 (Other: UW Madison); A536110 (Other: UW Madison)
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hip Preservation Surgery
Keywords: mindfulness; outcomes
MeSH Terms: interventions — Amyloid

STUDY DESIGN:
Intervention Model Description: single-blind, randomized controlled trial design
Who Masked: Care Provider
Masking Description: All healthcare providers involved in the care of the participant following surgery (surgeon, physician's assistants, nurses, medical assistants, etc.) will be blinded to the group assignment of each participant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Intervention plus Standard of Care (Experimental): The Foundations and Awareness modules of the HMP app require a minimum of 133 and 253 minutes, equating to less than 5 and less than 10 minutes per day on average, respectively. Date, duration, and content of usage will be recorded for each participant through the app. Participants will have access to the entire contents of the app for the full duration of the study.
  Interventions: Behavioral: Healthy Minds Program (HMP) App
- Standard of Care (No Intervention): Control group receives standard of care only

INTERVENTIONS:
Behavioral: Healthy Minds Program (HMP) App — The full HMP app includes 5 modules with practices designed to cultivate categories of mental and emotional skills linked to both hedonic and eudaimonic well-being. These include the cultivation of mindful attention (Awareness), positive relationships with self and others (Connection), insight into the nature of self and internal experience (Insight), and purpose, values, and meaning in life (Purpose), as well as an initial module which includes abbreviated introductions to the topics and lessons in all four areas (Foundations). For this study, the active intervention will include 4 weeks of training using the Foundations module followed by 4 weeks of training using the Awareness module.
  Arms: Mindfulness Intervention plus Standard of Care

SUMMARY:
Hip preservation surgery patients experience physical trauma, both in the physical injury itself and following surgery, and face potential long-lasting effects such as muscle weakness or diminished joint function, hip pain, and fear. Many of these patients report greater anxiety and depression following surgery, which can further compound negative outcomes in these patients. This study is a single-blind, randomized controlled trial design to evaluate the effects of a remotely-delivered 8-week mindfulness intervention on patient-reported outcomes following hip preservation surgery.

DETAILED DESCRIPTION:
The goal is to identify whether a mobile-based daily mindfulness program for the immediate eight weeks following hip preservation surgery improves outcomes in patients. The investigators hypothesize that patients who participate in a mindfulness intervention will have less pain, better hip function, greater quality of life, and improved scores on standardized patient reported outcome measures for 24 months following surgery.

The investigators expect their findings will re-direct post-operative strategies beyond the physical recovery in orthopedic surgery patients and improve long-term outcomes. To test the overall hypothesis and contribute significantly to understanding of the impact of a psychosocial intervention on outcomes in orthopedic surgery patients, the specific aim is to determine the influence of mindfulness training on patient-reported outcomes following hip preservation surgery.

* Specific Aim 1: To determine the influence of mindfulness training on patient-reported outcomes following hip preservation surgery

  * Hypothesis 1: Mindfulness training will be associated with improvements in pain, post-operative opiate use, hip function, quality of life and improved scores on standardized patient reported outcome measures for 24 months following hip preservation surgery
* Specific Aim 2: To determine the factors that influence mindfulness efficacy in patient-reported outcomes following hip preservation surgery

  * Hypothesis 2: Among participants in the mindfulness group, total duration of mindfulness training, female gender, and higher education level will be independently and positively associated with improvements in pain, hip function, and quality of life for 24 months following hip preservation surgery

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old at the time of the pre-operative visit
* Access to a mobile device compatible with the freely available Healthy Minds Program (HMP) App (Android or iOS)
* Participation in study 2019-0363

Exclusion Criteria:

* Prior diagnosis of serious mental illness (schizophrenia, bipolar disorder, schizoaffective disorder, etc).
* Significant prior experience with meditation or mindfulness, defined as greater than 30 minutes in a month during the past year

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in PROMIS Global Health Questionnaire (GHQ) Score | baseline, 3 months, 6 months, 12 months, 24 months
  Global quality of life (QoL) will be assessed via a 9-item questionnaire scored on a 0-100 scale where higher scores indicate better QoL, pain interference, and fatigue.
Change in PROMIS Anxiety and Depression Questionnaire Score | baseline, 3 months, 6 months, 12 months, 24 months
  Anxiety and depression will be assessed via an 8-item questionnaire scored from 0-5 where higher scores represents greater anxiety and depression.
Change in International Hip Outcome Tool (IHOT) Score | baseline, 3 months, 6 months, 12 months, 24 months
  Hip-related QoL is assessed via a 12-item survey scored from 0-10 where higher scores represent better hip-related quality of life.
Change in Modified Harris Hip Score (mHHS) | baseline, 3 months, 6 months, 12 months, 24 months
  Hip function is assessed via an 8-item survey scored on various scales with a total possible range of scores from 0-91 where higher scores indicate better hip pain and function.
Change in Single Assessment Numeric Evaluation (SANE) Score | baseline, 3 months, 6 months, 12 months, 24 months
  Current illness is assessed via a single item survey scored from 0-100 where a higher score represents closer to uninjured baseline.
Change in Hip Outcome Score (HOS-ADL and HOS-SS) | baseline, 3 months, 6 months, 12 months, 24 months
  Function with Activities of Daily Living and Sport Specific activities are assessed via a 28-items scored from 0-4 where higher scores indicate improved function.

SECONDARY OUTCOMES:
Total Duration of Mindfulness Training in the Mindfulness Group | up to 24 months
  The hypothesis is that among participants in the mindfulness group, total duration of mindfulness training, female gender, and higher education level will be independently and positively associated with improvements in pain, hip function, and quality of life for 24 months following hip preservation surgery.

OTHER OUTCOMES:
Summary of Pain Locations | baseline, 3 months, 6 months, 12 months, 24 months
  Pain location will be assessed by asking the participant to identify current location of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Watson, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No